CLINICAL TRIAL: NCT01957319
Title: Silybin Supplementation During HCV Therapy With Pegylated Interferon-α2b Plus Ribavirin Reduces Depression and Increases Work Ability
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Mariano Malaguarnera, Associate Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12/1997
Record Dates: First submitted 2013-09-25; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-09

CONDITIONS: Work Ability; Depression
MeSH Terms: conditions — Depression | interventions — Silybin; Vitamin E; Phospholipids; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Silybin - vitamin E - phospholipids complex (Active Comparator): Silybin 94 mg + vitamin E 90 mg + phospholipids 194 mg in one pill for 12 months.
  Interventions: Drug: Silybin 94 mg + vitamin E 90 mg + phospholipids 194 mg
- placebo (Placebo Comparator): sugar pill
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: Silybin 94 mg + vitamin E 90 mg + phospholipids 194 mg
  Arms: Silybin - vitamin E - phospholipids complex
Drug: sugar pill
  Arms: placebo

SUMMARY:
Background: Hepatitis C virus infection and interferon treatment have shown to be risk factors for depression, distressing, psychosocial burden and poor health-related quality of life.

Aim: To determine the effect of a Sylibin-vitamin E-phoshpolipids complex on work ability and whether health related factors (anxiety and depression) were associated with work ability in subjects with chronic hepatitis C treated with Peg-IFN-α and RBV.

Patients and Methods: In this prospective, randomized, placebo controlled, double blind clinical trial, 31 subjects (Group A) with chronic hepatitis, received Pegylated-Interferon-α2b (1.5 mg/kg per week) plus Ribavirin and placebo, while 31 subjects (Group B) received the same dosage of Pegylated-Interferon-α2b plus Ribavirin plus association of Silybin 94 mg + vitamin E 90 mg + phospholipids 194 mg in one pill for 12 months. All subjects underwent laboratory exams and questionnaires to evaluate depression (Beck Depression Inventory - BDI), anxiety (State-trait anxiety inventory - STAI) and work ability (Work ability Index - WAI).

ELIGIBILITY:
Inclusion Criteria:

* HCV infection

Exclusion Criteria:

* cancer severe jaundice pulmonary and renal chronic diseases prostatic diseases autoimmune diseases diabetes mellitus decompensated cirrhosis pregnancy hemoglobinopathies hemocromatosis

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Work ability index | 12 months
  Administration of questionnaire(Work ability Index - WAI)The work ability index is a tool to record the work ability of employees. It aims at identifying, at an early stage, health risks of early retirement an counteracting them. The questionnaire is aimed at: 1) the estimated current and future work ability; 2) diagnosed illness and the number of absenteeism days in the previous year; 3) the estimated sickness-related deterioration in the work performance; 4) mental ability reserves. The WAI evaluates current work ability compared with lifetime and in relation to the demands of the job, number of current diseases diagnosed by a physician, estimated work impairment due to diseases.

SECONDARY OUTCOMES:
depression | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Catania, Cannizzaro Hospital, Catania, Italy

REFERENCES:
- [Derived] Malaguarnera G, Bertino G, Chisari G, Motta M, Vecchio M, Vacante M, Caraci F, Greco C, Drago F, Nunnari G, Malaguarnera M. Silybin supplementation during HCV therapy with pegylated interferon-alpha plus ribavirin reduces depression and anxiety and increases work ability. BMC Psychiatry. 2016 Nov 15;16(1):398. doi: 10.1186/s12888-016-1115-z. PMID 27842532